CLINICAL TRIAL: NCT02349100
Title: Clinical Relevance of Positron Emission Tomography (PET) Imaging Following Endovascular Aneurysm Repair Using the Nellix Endoprosthesis
Brief Title: PET-CT After Nellix Implantation
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Michel Reijnen, M.D., PhD., Rijnstate Hospital
Other Study IDs: 1093
Record Dates: First submitted 2015-01-12; First posted 2015-01-28 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Aortic Aneurysm; Endovascular Repair
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treated group: Patient group treated with Nellix Endoprosthesis.
  Interventions: Device: Nellix Endoprosthesis

INTERVENTIONS:
Device: Nellix Endoprosthesis — Implantation of Nellix

SUMMARY:
To determine FDG uptake following uncomplicated EVAR using the Nellix endoprosthesis. Does uncomplicated EVAR using the nellix endoprosthesis result in increased FDG uptake and false positive PET imaging?

DETAILED DESCRIPTION:
One of the most devastating complications following endovascular aneurysm repair (EVAR) is infection of the used endoprosthesis. Because of the high mortality of secondary surgery following infection, patients with a possible endoprosthesis infection are treated using broadspectrum antibiotics during months, years or even life-long. Unfortunately, the diagnosis of an endoprosthesis infection is difficult and based upon clinical suspicion and non-specific symptoms (e.g. fever and weigth loss) only. Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) is often used as a diagnostic tool to identify infection following EVAR. Like infection, sterile physiologic inflammation following EVAR is also associated with increased metabolism and FDG uptake. This could result in (false-)positive PET imaging resulting in diagnostic errors and antibiotic overuse.

The Nellix endoprosthesis is a relatively new device used for EVAR. In present literature there is no data on the degree of physiologic inflammation following implantation of a Nellix device and the value of postoperative FDG-PET imaging to detect infection is not known. This makes the diagnosis of infection following Nellix implantation extremely difficult. This pilot is designed to determine physiologic FDG uptake following uncomplicated EVAR using the Nellix endoprosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with Nellix endoprosthesis

Exclusion Criteria:

* Diabetes Mellitus (Type 1 and type 2)
* Current known inflammation or malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with abdominal aortic aneurysms eligible for EVAS with Nellix endoprosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-07-13 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
Difference in physiological FDG uptake following Nellix EVAS implantation in patients without known infections or malignancies as measured by standard uptake values (SUV) | 1 month
  Comparing pre- and post-implantation FDG uptake with ROI set at the aneurysm and stent. Measured SUV from FDG emission will be compared and subtracted and the difference will be reported (in MBq/kg).

CONTACTS AND LOCATIONS:
Overall Officials: Michel Reijnen, PhD, MD, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate Ziekenhuis, Arnhem, Gelderland, Netherlands

REFERENCES:
- [Derived] Groot Jebbink E, van Den Ham LH, van Woudenberg BBJ, Slart RHJA, Zeebregts CJ, Rijnders TJM, Lardenoije JHP, Reijnen MMPJ. Physiological Appearance of Hybrid FDG-Positron Emission Tomography/Computed Tomography Imaging Following Uncomplicated Endovascular Aneurysm Sealing Using the Nellix Endoprosthesis. J Endovasc Ther. 2020 Jun;27(3):509-515. doi: 10.1177/1526602820913888. Epub 2020 Apr 15. PMID 32295455